CLINICAL TRIAL: NCT05484765
Title: The Effects of Smoking on Genotoxic and Histopathologic Damage in Exfoliated Oral Epithelial Cells and the Periodontium
Brief Title: Effects of Smoking on Oral Tissue Samples
Status: Completed | Type: Observational
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, Begum Alkan, Periodontology specialist, Istanbul Medipol University Hospital
Other Study IDs: ESGHDEOECP
Record Dates: First submitted 2022-07-01; First posted 2022-08-02 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Histopathology; Periodontitis; Smoking; Micronuclei
MeSH Terms: conditions — Periodontitis; Smoking

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Biospecimen Retention: Samples With DNA — smear samples, containing exfoliated oral epithelial cells, were taken from buccal and gingival mucosa
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Smoking negatively affects the prognosis of periodontal disease by impairing tissue healing. While micronucleus is the most popular parameter for demonstrating DNA damage, inflammatory cell and vascular densities are the most evaluated parameters for determining histopathologic changes in the periodontium. This cross-sectional study aimed to evaluate the effects of heavy cigarette smoking and generalized periodontitis on local genotoxic damage to exfoliated oral epithelial cells as well as histopathologic damage to the periodontium. The investigators hypothesized that the genotoxic and histopathologic damage would be increased in smokers with generalized periodontitis.

DETAILED DESCRIPTION:
Study design and Setting This was a single-center, investigator-blinded, cross-sectional study. Work was conducted at the Department of Periodontology in Istanbul, Turkey, between November 2018 and July 2019. The study procedure was conducted according to the guidelines of the Declaration of Helsinki and approved by the Ethics Committee of the university (Protocol code: 10840098-604.01.01-E.47596&10840098-604.01.01-E.4759; date of approval: 30 October 2018). Data from six non-smoking participants with healthy periodontium from our previous studies were used in this study as well. After the study was verbally explained to eligible subjects, those willing to participate signed a written, informed consent form. Personal, identifiable information about the subjects was kept confidential. The study was reviewed following the Strengthening the Reporting of Observational Studies in Epidemiology guidelines.

Participants Eighty systemically healthy subjects, both male and female, were enrolled in the study. Participants were recruited from patients who came to our department for periodontal examinations between November 2018 and July 2019. Diagnoses of clinically healthy periodontium and generalized periodontitis stages III-IV/grades B-C were performed according to the 2017 World Workshop on the Classification of Periodontal and Peri-implant Diseases and Conditions. Subjects were separated into four groups: smokers with generalized periodontitis (SGP; n = 20), non-smokers with generalized periodontitis (NGP; n = 20), smokers with clinically healthy periodontium (SHP; n = 20), and non-smokers with clinically healthy periodontium (NHP; n = 20). The following criteria needed to be met to be considered a periodontitis subject: the presence of generalized periodontitis, the presence of at least 20 teeth, the presence of a molar with an indication of gingivectomy, crown lengthening or extraction with a probing depth ≥ 5mm, clinical attachment loss ≥ 5 mm, and the presence of at least ten teeth with a probing depth ≥ 5 mm. The following criteria indicated a clinically healthy periodontium: a healthy and intact periodontium, no probing depth and bleeding on probing.

Clinical procedure All subjects answered a questionnaire that assessed age, gender, and educational level. A clinical evaluation of periodontal disease was conducted according to international standards. The CPPs, including plaque index, probing depth, bleeding on probing, and clinical attachment loss, were recorded from six sites per tooth from each subject using a periodontal probe by the same researcher. The sample collection and histopathologic evaluation procedures were performed as in our previous report. Briefly, smear samples were collected from the attached gingival mucosa of the upper premolar-molar area and the buccal mucosa of the matching cheek using two separate sterile cytobrushes. Samples were fixed on glass slides. Biopsy samples were taken from the vestibular area of the maxillary molars during tooth extraction or crown lengthening using a surgical blade and fixed in 10% formalin until analysis. During microscopic inspection, each subject rinsed their mouth before samples were obtained to reduce the possibility of artifacts through chromatin remainders.

Laboratory procedure To evaluate the exfoliated oral epithelial cells containing micronuclei counts (the primary outcome), the Feulgen reaction was performed on all smear samples. Cells were placed in a fixative for nuclear staining and analysis using Schiff's reagent. Micronuclei in the buccal and gingival smear samples were analyzed by observing them in oil immersion at 1000× magnification. One thousand cells were checked, and the count of micronuclei present was assessed. The occurrence of nuclear morphological changes, such as the presence of two nuclei within a cell, nuclei that appeared cinched with a Feulgen negative band, shrunken nuclei, condensed chromatin, nuclear disintegration involving the loss of nuclear integrity, and nuclear dissolution was estimated. A zigzag strategy was used to calculate the cells.

Histopathologic damage (the secondary outcome) was evaluated by focusing on inflammatory cell and vascular densities. Damage was assessed using a modified semi-quantitative histopathologic assessment method using a scale ranging from 0 to 3 (0: none, 1: mild, 2: moderate, and 3: intense). Tissue samples were fixed in paraffin wax, serially sectioned at a 4 µm thickness, stained with hematoxylin-eosin, and examined at 400× magnification. All smear and tissue samples were assayed concurrently and in the same laboratory by the same blinded investigator.

Bias The evaluation of each participant's systemic health status, dental history, and smoking habits was based on self-reported information regardless of official medical records. One researcher collected the data and samples from the participants while another researcher undertook the laboratory investigations. To avoid bias, five sample areas were randomly selected during the histologic examinations.

Study size The sample size was determined using G*Power version 3.1.9.4, assuming an alpha significance level of 0.05, a beta value of 0.1, and 90% power. As there were four study groups and a need for 20 participants per group, eighty subjects were included in the study.

Statistical methods The Number Cruncher Statistical System 2007 software program was used for all statistical analyses. Descriptive statistics (mean, standard deviation, median) were used to evaluate the data. The one-way analysis of variance test was used to compare the means of three or more normally distributed parameters. The Bonferroni test was used to determine the significant differences in pairwise comparisons between the groups. The Pearson chi-square test was used to compare qualitative data. Significance was evaluated at the p<0.01 and p<0.05 levels.

ELIGIBILITY:
Inclusion Criteria:

* Self-reporting as systemically healthy
* Aged between 18-65 years
* The presence of at least five teeth in each quadrant
* To need gingivectomy operations, crown lengthening procedures, or tooth extractions.
* Smokers had used cigarettes for at least five years with daily consumption of ≥ 20.

Exclusion Criteria:

* The presence of a known medical condition that could possibly bias the results
* Having a medical condition requiring antibiotic prophylaxis for dental treatment
* The presence of systemic medication taken within the previous six months
* Excessive alcohol consumption
* Currently undergoing nicotine replacement therapy
* Consuming tobacco products other than cigarettes
* Those with fixed orthodontic appliances
* History of periodontal therapy

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects were separated into four groups: smokers with generalized periodontitis (SGP; n = 20), non-smokers with generalized periodontitis (NGP; n = 20), smokers with clinically healthy periodontium (SHP; n = 20), and non-smokers with clinically healthy periodontium (NHP; n = 20). The following criteria needed to be met to be considered a periodontitis subject: the presence of generalized periodontitis, the presence of at least 20 teeth, the presence of a molar with an indication of gingivectomy, crown lengthening or extraction with a PD ≥ 5mm, clinical attachment loss ≥ 5 mm, and the presence of at least ten teeth with a PD ≥ 5 mm. The following criteria indicated a clinically healthy periodontium: a healthy and intact periodontium, no PD and BOP.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-07-15 (Actual); Study Completion 2019-07-20 (Actual)

PRIMARY OUTCOMES:
Micronuclei counts | 1 year
  During mitosis, loss of chromatin from chromosomal DNA is manifested by extra-small, abnormal nuclear structures called micronuclei. Of the available cytogenetic analyses, the micronucleus assay is one of the most popular methods for detecting structural and numerical nuclear abnormalities due to its reliability and simplicity. This genotoxic biomonitoring assay makes it possible to provide evidence for the biological assessment of disease susceptibility, diagnosis, and staging in subjects exposed to environmental risk factors.Briefly, smear samples were collected from the attached gingival mucosa of the upper premolar-molar area and the buccal mucosa of the matching cheek using two separate sterile cytobrushes. Samples were fixed on glass slides.
Histopathologic changes | 1 year
  Histopathologic damage was evaluated by focusing on inflammatory cell and vascular densities.Biopsy samples were taken from the vestibular area of the maxillary molars during tooth extraction or crown lengthening using a 15C surgical blade and fixed in 10% formalin until analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Begum Alkan, Principal Investigator — Private Practice of Periodontology (formerly Istanbul Medipol University)
Locations (1):
- Begüm Alkan, Istanbul, Turkey (Türkiye)